CLINICAL TRIAL: NCT02167334
Title: Non Invasive Ventilation (NIV) Versus Spontaneous Breathing for Preoxygenation During Ear, Nose, and Throat (ENT) Panendoscopy. A Controlled, Prospective, Randomized Study.
Brief Title: Using Positive Pressure Ventilation for Preoxygenation During Panendoscopy.
Acronym: PANNIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI12-DR-DIMOV; 2012-A01053-40 (Other: ID-RCB)
Record Dates: First submitted 2014-06-11; First posted 2014-06-19 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: ENT Cancer Screening
Keywords: panendoscopy; preoxygenation; non invasive ventilation
MeSH Terms: interventions — Positive-Pressure Respiration; Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- positive pressure ventilation (Experimental): Positive Pressure Ventilation with a 4 cmH2O inhale pressure, a positive end-expiratory pressure of 4 cm H2O, a trigger 2, an inspiratory slope of 0, an inhaled oxygen fraction of 100% administered at a 10 L / min flow.
  Interventions: Device: positive pressure ventilation
- Oxygenation with simple breathing mask (Active Comparator): spontaneously breathing preoxygenation with adapted face mask, to restrict leakage, at 10L/min oxygen, with inhaled fraction of 100% and a 2 L balloon volume.
  Interventions: Procedure: Oxygenation with simple breathing mask

INTERVENTIONS:
Device: positive pressure ventilation — Positive Pressure Ventilation with a 4 cmH2O inhale pressure, a positive end-expiratory pressure of 4 cm H2O, a trigger 2, an inspiratory slope of 0, an inhaled oxygen fraction of 100% administered at a 10 L / min flow.
  Other Names: non invasive ventilation (NIV)
  Arms: positive pressure ventilation
Procedure: Oxygenation with simple breathing mask — Spontaneously breathing preoxygenation with adapted face mask, to restrict leakage, at 10L/min oxygen, with inhaled fraction of 100% and a 2 L balloon volume.
  Arms: Oxygenation with simple breathing mask

SUMMARY:
the aim of the study is to determine if Spontaneous Ventilation with Positive Pressure Ventilation (PPV) preoxygenation allows a longer non hypoxemic apnea time during panendoscopy compared to spontaneous breathing preoxygenation.

the hypothesis is PPV extends the residual functional capacity of lung so it provides more oxygen during apnea.

ELIGIBILITY:
Inclusion Criteria:

* patient going for scheduled panendoscopy under general anesthesia

Exclusion Criteria:

* BMI upper to 35 kg/m2
* pregnancy
* requirement of jet ventilation
* tracheostomy
* acute respiratory failure: pneumonia, pulmonary embolism
* health insurance careless

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-09; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
non hypoxemic apnea time | up to 5 minutes after stopping oxygenation
  time the oxygen saturation is going down to 90% during apnea

SECONDARY OUTCOMES:
surgical laryngoscopy frequency | up to 15 minutes after stopping oxygenation
  number of stopped surgical laryngoscopy because of a low oxygen saturation under 90% with necessity to ventilate the patients during apnea
preoxygenation time | up to 10 min after the start of oxygenation
  time to reach expired oxygen fraction to 90%

CONTACTS AND LOCATIONS:
Overall Officials: Osama ABOU ARAB, MD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France

REFERENCES:
- [Result] Abou-Arab O, Guinot PG, Dimov E, Diouf M, de Broca B, Biet A, Zaatar R, Bernard E, Dupont H, Lorne E. Low-positive pressure ventilation improves non-hypoxaemic apnoea tolerance during ear, nose and throat pan-endoscopy: A randomised controlled trial. Eur J Anaesthesiol. 2016 Apr;33(4):269-74. doi: 10.1097/EJA.0000000000000394. PMID 26716862